CLINICAL TRIAL: NCT02702362
Title: Repeated Stimulation of the Precuneus in Chronic Patients in Minimally Conscious State: a Placebo-controlled Randomized Clinical Trial
Brief Title: tDCS on Precuneus in MCS: Repeated Stimulations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Wangshan Huang, graduate student, Hangzhou Normal University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/302/A
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Patients in Minimally Conscious State After a Severe Brain Injury
Keywords: disorders of consciousness; minimally conscious state; traumatic brain injury; stroke; transcranial direct current stimulation
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Brain Injuries, Traumatic; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anodal stimulation (Active Comparator): Patients received anodal tDCS (on the precuneus ) every day for 5 days (tDCS of 2mA during 20minutes). A CRS-R is performed at baseline (before the first stimulation) and after each tDCS.
  A final CRS-R is performed 5 days after the end of the session to assess the potential long term effects of the tDCS.
  Interventions: Device: transcranial direct current stimulation
- sham stimulation (Sham Comparator): Patients received sham tDCS (5 secondes of stimulation) every day for 5 days. A CRS-R is performed at baseline (before the first stimulation) and after each tDCS. A final CRS-R is performed 5 days after the end of the session.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — anodal transcranial direct current stimulation on the precuneus cortex for the anodal session and sham stimulation (5secondes of tDCS) for the sham session.

SUMMARY:
In this study researchers will apply transcranial direct current stimulation (tDCS) for 5 consecutive days in chronic patients in minimally conscious state (MCS).

DETAILED DESCRIPTION:
Positive effects of tDCS in patients in MCS was showed in a recent study published in Neurology. But the effects went down after 1 or 2 hours. To increase the lasting of the effects, a new study will evaluate the effects of tDCS on the precuneus cortex for 5 consecutive days in chronic patients in MCS.

2 sessions of 5 days of stimulation will be realized, one session will be real (anodal stimulation) and one placebo (sham stimulation). After each stimulation, behavioral improvement will be assessed with the Coma Recovery Scale Revised (CRS-R). A final assessment will be done 5 days after the end of the sessions to assess the long term effect of the tDCS.

Researchers expected to see an improvement of the CRS-R total score at the end of the anodal session and that this improvement persists for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* post comatose patients
* patients in minimally conscious state
* patients with stable condition
* patients free of sedative drugs and Na+ or Ca++ blockers (e.g., carbamazepine) or NMDA receptor antagonist (e.g., dextromethorphan)

Exclusion Criteria:

* premorbid neurology antecedent
* patients in coma or vegetative state
* patients < 1 months after the acute brain injury
* patients with a metallic cerebral implant or a pacemaker (in line with the safety criteria for tDCS in humans)

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in the CRS-R total score | After each stimulation and 5 days later for anodal and sham sessions (total: 1 month)
  Improvement of the CRS-R total score after the end of the anodal session and 5 days later but no change for the sham session

SECONDARY OUTCOMES:
Influence of the time since insult | one month
  Influence of the time since insult of the results. Researchers expected that the longer a patient is in MCS, the lower is his/her improvement after the tDCS session.